CLINICAL TRIAL: NCT06935019
Title: TRIAGE-GS: A Randomized Controlled Trial of a Genomics-first Approach to Rare Disease Diagnosis
Brief Title: TRIAGE-GS: Towards Reducing Inefficiencies Affecting Genetics Encounters Through Genome Sequencing
Acronym: TRIAGE-GS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Children's Hospital of Eastern Ontario (Other); Toronto Metropolitan University (Other)
Responsible Party: Principal Investigator, Gregory Costain, Staff Physician, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CTO5061
Record Dates: First submitted 2025-03-28; First posted 2025-04-18 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Genetic Conditions
Keywords: TRIAGE-GS

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GS-first arm (Experimental): The intervention is receiving immediate clinical routine GS, prior to evaluation by a medical geneticist. Pre-test counselling will be done by a research genetic counsellor. Results of GS will be returned during the participant's first visit to Genetics Clinic by their clinical team. Subsequent clinical care (including any other clinically indicated genetic testing or workup) will be arranged by the medical geneticist in clinic.
  Interventions: Genetic: Genome sequencing pre-geneticist evaluation
- Standard-of-care arm (No Intervention): The intervention group will be compared to the standard-of-care group, where evaluation by a medical geneticist in Genetics Clinic is a prerequisite to ordering of genetic testing. Clinical workups and genetic testing are ordered at the discretion of the medical geneticist involved in their clinical care, following evaluation.

INTERVENTIONS:
Genetic: Genome sequencing pre-geneticist evaluation — The intervention is receiving immediate clinical routine GS, prior to evaluation by a medical geneticist. Pre-test counselling will be done by a research genetic counsellor. Results of GS will be returned during the participant's first visit to Genetics Clinic by their clinical team. Subsequent clinical care (including any other clinically indicated genetic testing or workup) will be arranged by the medical geneticist in clinic.
  Arms: GS-first arm

SUMMARY:
Individually rare genetic diseases are collectively common, and affect many Canadian families. Making the right diagnosis is both important and challenging. Healthcare providers and families often remain in the dark for too long, limited by the scope and speed of current genetic testing.

The goal of this clinical trial is to learn if performing genome sequencing (a comprehensive genetic test) as soon as a rare genetic disease is suspected is more effective than usual care, where a person waits to see a genetics specialist and then typically gets offered more targeted testing. Researchers will compare a "genome-sequencing first" approach to the standard-of-care in individuals who were referred to the Genetics Clinic at either SickKids or CHEO and recently had their referral accepted by the clinic.

The main questions this clinical trial aims to answer are:

1. Are there more and faster diagnoses with a "genome sequencing first" approach compared to standard-of-care?
2. What do patients, families, and healthcare providers think about a "genome sequencing first" approach compared to standard-of-care?
3. What is the financial impact of a "genome sequencing first" approach compared to standard-of-care on the healthcare system?

Participants will be asked to:

* Let us review their medical records.
* Complete up to 5 questionnaires over the course of the study.
* Give a blood sample for clinical genome sequencing (if in the genome sequencing first group).

This study aims to provide the robust evidence needed to improve care pathways for rare disease diagnosis in Canada. The findings also promise to help translate new genetic technologies into the clinic. Earlier diagnosis is a key first step towards personalized care, targeted treatments, and better outcomes.

DETAILED DESCRIPTION:
This is a multi-centre, prospective, interventional, open randomized controlled trial that compares patient outcomes generated by clinical whole genome sequencing (GS) initiated at time of referral triage (i.e., prior to evaluation with a medical geneticist) to standard-of-care, where genetic testing is ordered post-evaluation. 200 individuals referred to SickKids or CHEO for suspected undiagnosed rare disease (RD) will be enrolled, along with their biological parents when possible. The purpose of this study is to examine the safety, utility, and feasibility of a "genomics first" diagnostic pathway for RD. The investigators hypothesize that a GS-first pathway will have non-inferior diagnostic yield and lead to a shorter duration of time to RD diagnosis, fewer diagnostics-focused clinic visits, and improved stakeholder satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Referral accepted to the Genetics Clinic at SickKids or CHEO within 7 days of screening for study eligibility.
* Referral is for a patient that is ≤18 years old.
* Reason for referral is a suspected but as-yet-undiagnosed RD
* A genetic aetiology is a possible explanation for the phenotype such that genetic testing is likely to be offered in Genetics Clinic, as determined by the research team.

Exclusion Criteria:

* Patient has a known or suspected clinical diagnosis using established criteria of a genetic condition with low locus heterogeneity (e.g., HHT, fCCM, NF1, TSC, others)
* Referral considered "Urgent" using established site criteria.
* Genome-wide sequencing (exome sequencing or GS) or a comprehensive panel that encompasses all genes relevant for the reported phenotype previously completed on a clinical or research basis.
* Patient or family member previously assessed by a medical geneticist within the last 2 years for the same phenotype(s).
* Patient lacks Ontario Health Insurance Plan (OHIP) or comparable coverage (as this will limit options for standard genetic testing).
* Referral is solely to facilitate familial variant testing or for genetic counselling.
* A family member is already enrolled in the study and was referred for the same indication.
* Patient/family does not provide informed consent to participate within 2 weeks of being approached.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-05-14 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Determine the time-to-event (diagnosis or no active follow-up) of a GS-first (pre-geneticist evaluation) outpatient care model for rare disease compared to standard of care. | From date of randomization until the date of the disclosure of diagnosis/plan, up to 18 months.
  The primary outcome measure for Aim 1 is a time-to-event variable. The event of interest is "diagnosis or no active follow-up," as measured for each participant from the date of randomization to the date of disclosure of the diagnosis/plan. Selection of a composite event variable was based on input from patients, families, and clinicians regarding the utility of negative GS results in certain scenarios. For example, a negative GS result might lower the index of suspicion for Mendelian disorders of known genetic basis, such that no further testing or short-term follow-up is recommended, or a clinical diagnosis of exclusion is made with confidence.
Compare clinical utility of GS-first to standard of care from the perspectives of care teams. | 0-2 weeks after the first results disclosure to the participant/family.
  The main outcome for Aim 2 will be differences in C-GUIDE total score, comparing the perceived utility of GS (in the GS-first group) with the first genetic test initiated by the geneticist for participants in the standard-of-care group.
Compare personal utility of GS-first to standard-of-care from the perspectives of patients, families, and care teams. | 0-2 weeks after the first results disclosure to the participant/family.
  The other main outcome for Aim 2 will be differences in GENE-U total score, comparing the perceived utility of GS (in the GS-first group) with the first genetic test initiated by the geneticist for participants in the standard-of-care group.
Assess cost-effectiveness as the incremental cost per additional case detected for GS-first compared to standard-of-care from a healthcare system payer perspective. | Overall during the study period (up to 18 months).
  An incremental cost-effectiveness analysis (CEA) that compares GS-first to standard-of-care per additional positive finding will be undertaken from the perspectives of the healthcare system and society. The economic evaluation will use recommended methods.

SECONDARY OUTCOMES:
Primary diagnostic yield | Overall during the study period (up to 18 months), and within a 6-month time interval from the date of randomization.
Proportion of participants with dual diagnoses | Overall during the study period (up to 18 months).
Proportion of participants with partial genetic diagnoses | Overall during the study period (up to 18 months).
Proportion of participants with potential genetic diagnoses | Overall during the study period (up to 18 months).
Proportion of participants with variants of uncertain significance deemed non-contributory by the clinician | Overall during the study period (up to 18 months).
Proportion of participants with secondary/incidental findings | Overall during the study period (up to 18 months).
Number of new informative HPO terms coded after evaluation by a geneticist (compared with data extracted from collateral records at the time of the referral) | Overall during the study period (up to 18 months).
  This can be stratified by the original referral source (i.e., internal referrals from providers at SickKids/CHEO vs. referrals from external providers).
Differences in amount of time/effort required for reporting genome sequencing | Overall during the study period (up to 18 months).
  Including time recorded by the analyst, number/type of variants unnecessarily reported due to incomplete phenotypic information, etc.
Number of diagnoses missed by GS in the intervention arm that were later made after geneticist evaluation | Overall during the study period (up to 18 months).
  Including variants seen by GS that were not reported based on phenotypic information known prior to geneticist assessment, variants identified on reanalysis using new HPO terms entered post-geneticist assessment, or variant types (e.g., repeat expansions) that were missed by GS due to technical limitations, etc.
Incremental cost per unit improvement in C-GUIDE score | Overall during the study period (up to 18 months).
  A secondary analysis under the CEA will examine the incremental cost per unit improvement in C-GUIDE score

OTHER OUTCOMES:
Motivations and barriers to study participation | 0-2 weeks post-study enrolment, or offered immediately after declining to participate.
  The investigators will assess factors that motivated families to participate, as well as factors that presented potential barriers at T0. These questions were developed by the study team for the purposes of this study. This component of the outcome measures will also be offered to individuals who decline to participate in an attempt to better understand barriers and improve the study.
Sociodemographics | 0-2 weeks post-study enrolment.
  The study team will collect detailed sociodemographic, and equity related variables at T0. Some of this information is already collected in the electronic medical record as part of routine clinic visits. In cases where this information is readily available, the study team will gather it from the chart and not ask families to answer the questions again.
BRIEF Health Literacy Screening Tool | 0-2 weeks post-study enrolment.
  Health literacy is described as the degree to which one can read, understand, exchange, and use health information and resources. The BRIEF: Health Literacy Screening Tool consists of four questions that participants respond to on a 5-point Likert scale, and will be administered at T0. It measures patients' health literacy, where higher scores indicate higher levels of health literacy.
Everyday Discrimination Scale (Short Version) | 0-2 weeks post-study enrolment.
  The Everyday Discrimination Scale (Short Version) consists of 6 items intended to capture respondents' experiences with discrimination in their life. It is reliable (α = 0.77). It will be administered at T0 only.
University of North Carolina Genomic Knowledge Scale (UNC-GKS) | 0-2 weeks after study enrolment; 0-2 weeks after pre-test counselling; 0-2 weeks after each results disclosure (up to a maximum of 3 disclosures).
  The UNC-GKS consists of 25 items to measure genomic knowledge among people facing decisions about genome-wide sequencing. It was shown to assess genomic knowledge with good internal reliability (Cronbach's α = 0.90), and convergent validity supported by association with health literacy and numeracy (rs = 0.41-0.46). It will be administered at T0, T1, T2 and TN (up to a maximum of T4) to allow comparison throughout families' diagnostic journeys, and assess whether there are differences in knowledge/understanding between the study arms.
Short-Form State-Trait Anxiety Inventory (STAI) | 0-2 weeks after study enrolment; 0-2 weeks after pre-test counselling; 0-2 weeks after each results disclosure (up to a maximum of 3 disclosures).
  The short form of the Spielberger STAI consists of 6 items that measure fluctuations in state anxiety.60 This short form version was found to be reliable (α = 0.32) and valid as compared to the full (20-item) version.60 It will be administered at all time points, starting at T0.
Genetic Counselling Satisfaction Scale (GCSS) | 0-2 weeks after pre-test counselling; 0-2 weeks after each results disclosure (up to a maximum of 3 disclosures).
  The GCSS is a 6-item instrument to measure an individual's satisfaction with the genetic counselling they received. It is reliable (Cronbach's α = 0.90) and described as face valid. It will be administered at all time points, starting at T1.
GENEtic Utility (GENE-U) Scale for Pediatric Diagnostic Testing | 0-2 weeks after each results disclosure (up to a maximum of 3 disclosures).
  The GENEtic Utility (GENE-U) scale consists of 21 items that capture the caregiver's test-specific reactions. It is designed for administration after test completion and results disclosure, and it is intended to be complementary to assessments of clinical utility. Convergent validity has been calculated using the Pearson correlation coefficient between scores on the GENE-U and measures of theoretically related constructs, and scores supported construct validity. It will be administered at all time points, starting at T2.
Clinician-reported Genetic Testing Utility InDEx (C-GUIDE™) | 0-2 weeks after each results disclosure.
  To capture clinicians' assessment of utility, the investigators will use the Clinician-reported Genetic Testing Utility InDEx (C-GUIDE™). C-GUIDE™ was developed to assess the post-test utility of diagnostic and secondary variants generated by germline genetic tests. Evaluation using case vignettes has demonstrated that C-GUIDE v1.2 is reliable (Krippendorff's α=0.675) and valid. Consulting geneticists or genetic counsellors will be asked to complete C-GUIDE™ ratings on each enrolled index case within two weeks of the first result disclosure (T1), and for each subsequent result disclosure during the study period (TN), to allow for an assessment of clinical utility overtime.
Supplemental aspects of clinical utility | 0-2 weeks after each results disclosure.
  The study team will supplement the C-GUIDE™ ratings by documenting information from the patient's chart about the care plan that was recommended based each result (e.g., follow-up visits, referrals, surveillance plans, investigations, treatments, procedures). The source for this information will be the consult note written by the consulting geneticist following results disclosure.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - The Hospital for Sick Children, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Study protocol, including statistical analysis plan, and informed consent form template will be submitted for open-access publication. Individual participant data can be shared upon request and execution of a data transfer agreement when consent was given by the participant or their substitute decision maker. Potentially identifying data (e.g., variable represented less than 5 times in the cohort) will not be shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be made available within 6 months of the study's conclusion, and will remain available for at least 5 years.
Access Criteria: Accessing the data set will require a signed data transfer agreement.
URL: https://triage-gs.ca/

REFERENCES:
- [Derived] Stanley KJ, Chisholm C, Gillespie MK, Caluseriu O, Del Signore N, Elango S, Hartley T, Hewson S, Kim RH, McSheffrey G, Mendoza-Londono R, Sawyer SL, Somerville M, Venkataramanan V, White-Brown A, Telesca S, Shickh S, Marshall CR, Ungar WJ, Hayeems RZ, Bhawra J, Boycott KM, Costain G. TRIAGE-GS: protocol for a randomised controlled trial of a genomics-first approach to rare disease diagnosis for patients awaiting assessment by a clinical geneticist. BMJ Open. 2025 Aug 10;15(8):e107603. doi: 10.1136/bmjopen-2025-107603. PMID 40784761